CLINICAL TRIAL: NCT04022525
Title: Assessment of Leflunomide Efficacy and Hepatotoxicity in Patients With Rheumatoid Arthritis Through Pharmacokinetic and Genetic Approaches
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Abdelkhalik Ahmed Mohamed, Principal Investigator, Assiut University
Other Study IDs: 2016/12/28-006
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- leflunomide responsive vs non-responsive
  Interventions: Drug: Leflunomide 20Mg Tab

INTERVENTIONS:
Drug: Leflunomide 20Mg Tab — blood samples of rheumatoid patients will be collected for SNPs detection and drug assay

SUMMARY:
The RA patients receiving leflunomide for more than one month, and not receiving other DMARDs (except hydroxychloroquine), will be enrolled to assess their disease activity. Blood samples will be collected for genetic studies and pharmacokinetic assay of the blood levels of the drug and its active metabolite.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients already receiving leflunomide with or without Hydroxychloroquine but without other Disease modifying agents

Exclusion Criteria:

* Those diagnosed with other rheumatic diseases or Rheumatoid patients receiving disease modifying agents other than leflunomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients from both sexes with different disease activity status receiving solely leflunomide with or without hydroxychloroquine
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of single nucleotide polymorphisms associated with response to the drug | one -two years
  SNPs associated with the response or adverse drug reactions will be detected and correlated with the ratio of leflunomide to its active metabolite

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt